CLINICAL TRIAL: NCT05478278
Title: A Phase 1, Two-Part Study in Healthy Volunteers to Evaluate The Effect of Psilocybin on Cardiac Repolarization and The Effect of Food on Psilocybin Pharmacokinetics
Brief Title: An Evaluation of Psilocybin's Effect on Cardiac Repolarization and the Effect of Food on Psilocybin's Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Usona Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PSIL102-TQT
Record Dates: First submitted 2022-07-14; First posted 2022-07-28 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: QTc Interval; Pharmacokinetics
Keywords: Psilocybin, Psychedelics
MeSH Terms: interventions — Psilocybin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Treatment A (IP at Therapeutic Dose) (Experimental): A single therapeutic dose of psilocybin.
  Interventions: Drug: Psilocybin
- Part 1: Treatment B (IP at Supratherapeutic Dose) (Experimental): A single supratherapeutic dose of psilocybin.
  Interventions: Drug: Psilocybin
- Part 1: Treatment C (Placebo - Negative Control) (Placebo Comparator): A single dose of placebo-to-match psilocybin MCC capsules.
  Interventions: Drug: Micro-Crystalline Cellulose
- Part 1: Treatment D (Placebo - Positive Control) (Active Comparator): A single 400 mg dose of moxifloxacin.
  Interventions: Drug: Moxifloxacin
- Part 2: IP at Therapeutic Dose (Fasted Conditions) (Experimental): A single therapeutic dose of psilocybin administered under fasted conditions.
  Interventions: Drug: Psilocybin
- Part 2: IP at Therapeutic Dose (Fed Conditions) (Experimental): A single therapeutic dose of psilocybin under fed conditions.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — The psilocybin used in this study is synthetically manufactured in a laboratory and meets quality specifications suitable for human research use. The active drug is encapsulated using a hydroxypropyl methylcellulose (HPMC) capsule and contains psilocybin (API only in a capsule).
  Other Names: Psilocybine; Psilocibin; Indocybin
  Arms: Part 1: Treatment A (IP at Therapeutic Dose); Part 1: Treatment B (IP at Supratherapeutic Dose); Part 2: IP at Therapeutic Dose (Fasted Conditions); Part 2: IP at Therapeutic Dose (Fed Conditions)
Drug: Moxifloxacin — The positive comparator used in this study is a 400 mg moxifloxacin tablet.
  Other Names: Avelox; Moxeza
  Arms: Part 1: Treatment D (Placebo - Positive Control)
Drug: Micro-Crystalline Cellulose — The placebo used in this study is encapsulated using a HPMC capsule and contains micro-crystalline cellulose.
  Arms: Part 1: Treatment C (Placebo - Negative Control)

SUMMARY:
This study is comprised of two parts. The purpose of the first part of this study is to evaluate the effects of a supratherapeutic dose of psilocybin on cardiac repolarization. The purpose of the second part of the study is to evaluate the effects of food on the pharmacokinetics of psilocybin.

DETAILED DESCRIPTION:
Part one of this study will be a double-blind, single-dose, randomized, placebo-controlled, 4-treatment, 4-period, 12-sequence crossover design in 36 healthy volunteers (adult male and/or female subjects). Subjects will be randomly assigned to 1 of 12 different treatment administration sequences, whereby each sequence will include 3 double-blind treatments (therapeutic dose of psilocybin, supratherapeutic dose of psilocybin, and placebo) and 1 open-label positive control treatment (moxifloxacin).

Part two of this study will be an open-label, randomized, 2-period, 2-sequence crossover design in 24 healthy volunteers (adult male and/or female subjects). Each assigned treatment will be administered under fasting or fed conditions as a single dose on Day 1 of the respective study period.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form (ICF)
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Healthy adult male or female
* Aged at least 18 years but not older than 65 years, inclusive
* Body mass index (BMI) within 18.0 kg/m2 to 32.0 kg/m2 (for Part 1) or to 33.0 kg/m2 (for Part 2), inclusively

Exclusion Criteria:

* History of significant hypersensitivity to psilocybin or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability
* History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
* Showing suicidal ideation or behavior as per the Columbia Suicide Severity Rating Scale (C-SSRS) administered at screening
* Presence of out-of-range cardiac interval (PR < 110 msec, PR > 200 msec, QRS < 60 msec, QRS >110 msec and QTcF > 450 msec for males and > 470 for females) on the ECG at screening or other clinically significant ECG abnormalities, unless deemed non-significant by an Investigator
* History of risk factors for Torsades de Pointes (TdP), including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, angina, or clinically significant abnormal laboratory assessments including hypokalemia, hypercalcemia, or hypomagnesaemia
* Family history of long QT syndrome or Brugada syndrome
* Any clinically significant illness in the 28 days prior to the first study drug administration
* Intake of psilocybin or any other psychedelic (including 3,4-methylenedioxymethamphetamine [MDMA] and ketamine) in the 28 days prior to the first study drug administration
* Not suitable for participation in the study at the discretion of the Principal Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Part 1: Change from baseline (Day -1) QTcF (ΔΔQTcF) following up to 24 hours post administration of a supratherapeutic dose of psilocybin. | Up to 24 hours post-dose
  Replicate electrocardiograms (ECGs) (10 ECG replicates) for the determination of ΔQTc interval will be extracted from the continuous digital 12-lead ECG recording at the -0.75, -0.50, and -0.25 hours prior to dosing and then at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose.
Part 2: Change from baseline (T=0 hours) of AUC of psilocybin and its metabolite psilocin following up to 24 hours post administration of a therapeutic dose of psilocybin under fed and fasted conditions. | Up to 24 hours post-dose
  Pharmacokinetic endpoints for psilocybin and psilocin (AUC) will be evaluated at 0.00, 0.25, 0.50, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose.
Part 2: Change from baseline (T=0 hours) of Cmax of psilocybin and its metabolite psilocin following up to 24 hours post administration of a therapeutic dose of psilocybin under fed and fasted conditions. | Up to 24 hours post-dose
  Pharmacokinetic endpoints for psilocybin and psilocin (CMax) will be evaluated at 0.00, 0.25, 0.50, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose.
Part 2: Change from baseline (T=0 hours) of Tmax of psilocybin and its metabolite psilocin following up to 24 hours post administration of a therapeutic dose of psilocybin under fed and fasted conditions. | Up to 24 hours post-dose
  Pharmacokinetic endpoints for psilocybin and psilocin (TMax) will be evaluated at 0.00, 0.25, 0.50, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose.

SECONDARY OUTCOMES:
Part 1: Number of participants with Treatment-Related Adverse Events as assessed by CTCAE v4.0. | Up to 30 Days Post Dose
  Number of participants with TEAEs following administration of psilocybin and moxifloxacin.
Part 2: Number of participants with Treatment-Related Adverse Events as assessed by CTCAE v4.0 | Up to 15 Days Post Dose
  Number of participants with TEAE following administration of psilocybin.

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Clinical Kansas, Inc, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carhart-Harris RL, Leech R, Hellyer PJ, Shanahan M, Feilding A, Tagliazucchi E, Chialvo DR, Nutt D. The entropic brain: a theory of conscious states informed by neuroimaging research with psychedelic drugs. Front Hum Neurosci. 2014 Feb 3;8:20. doi: 10.3389/fnhum.2014.00020. eCollection 2014. PMID 24550805
- [Background] Nichols DE. Hallucinogens. Pharmacol Ther. 2004 Feb;101(2):131-81. doi: 10.1016/j.pharmthera.2003.11.002. PMID 14761703
- [Background] Passie T, Seifert J, Schneider U, Emrich HM. The pharmacology of psilocybin. Addict Biol. 2002 Oct;7(4):357-64. doi: 10.1080/1355621021000005937. PMID 14578010
- [Background] Carhart-Harris RL, Nutt DJ. Experienced drug users assess the relative harms and benefits of drugs: a web-based survey. J Psychoactive Drugs. 2013 Sep-Oct;45(4):322-8. doi: 10.1080/02791072.2013.825034. PMID 24377171
- [Background] Nutt DJ, King LA, Phillips LD; Independent Scientific Committee on Drugs. Drug harms in the UK: a multicriteria decision analysis. Lancet. 2010 Nov 6;376(9752):1558-65. doi: 10.1016/S0140-6736(10)61462-6. Epub 2010 Oct 29. PMID 21036393
- [Background] Hasler F, Bourquin D, Brenneisen R, Bar T, Vollenweider FX. Determination of psilocin and 4-hydroxyindole-3-acetic acid in plasma by HPLC-ECD and pharmacokinetic profiles of oral and intravenous psilocybin in man. Pharm Acta Helv. 1997 Jun;72(3):175-84. doi: 10.1016/s0031-6865(97)00014-9. PMID 9204776
- [Background] Brown RT, Nicholas CR, Cozzi NV, Gassman MC, Cooper KM, Muller D, Thomas CD, Hetzel SJ, Henriquez KM, Ribaudo AS, Hutson PR. Pharmacokinetics of Escalating Doses of Oral Psilocybin in Healthy Adults. Clin Pharmacokinet. 2017 Dec;56(12):1543-1554. doi: 10.1007/s40262-017-0540-6. PMID 28353056
- [Background] Madsen MK, Fisher PM, Burmester D, Dyssegaard A, Stenbaek DS, Kristiansen S, Johansen SS, Lehel S, Linnet K, Svarer C, Erritzoe D, Ozenne B, Knudsen GM. Psychedelic effects of psilocybin correlate with serotonin 2A receptor occupancy and plasma psilocin levels. Neuropsychopharmacology. 2019 Jun;44(7):1328-1334. doi: 10.1038/s41386-019-0324-9. Epub 2019 Jan 26. PMID 30685771
- [Background] Manevski N, Kurkela M, Hoglund C, Mauriala T, Court MH, Yli-Kauhaluoma J, Finel M. Glucuronidation of psilocin and 4-hydroxyindole by the human UDP-glucuronosyltransferases. Drug Metab Dispos. 2010 Mar;38(3):386-95. doi: 10.1124/dmd.109.031138. Epub 2009 Dec 10. PMID 20007669
- [Background] Hasler F, Bourquin D, Brenneisen R, Vollenweider FX. Renal excretion profiles of psilocin following oral administration of psilocybin: a controlled study in man. J Pharm Biomed Anal. 2002 Sep 5;30(2):331-9. doi: 10.1016/s0731-7085(02)00278-9. PMID 12191719
- [Background] Darpo B, Benson C, Dota C, Ferber G, Garnett C, Green CL, Jarugula V, Johannesen L, Keirns J, Krudys K, Liu J, Ortemann-Renon C, Riley S, Sarapa N, Smith B, Stoltz RR, Zhou M, Stockbridge N. Results from the IQ-CSRC prospective study support replacement of the thorough QT study by QT assessment in the early clinical phase. Clin Pharmacol Ther. 2015 Apr;97(4):326-35. doi: 10.1002/cpt.60. PMID 25670536
- [Background] Ferber G, Zhou M, Darpo B. Detection of QTc effects in small studies--implications for replacing the thorough QT study. Ann Noninvasive Electrocardiol. 2015 Jul;20(4):368-77. doi: 10.1111/anec.12227. Epub 2014 Nov 4. PMID 25367715
- [Background] Huang DP, Chen J, Dang Q, Tsong Y. Assay sensitivity in "Hybrid thorough QT/QTc (TQT)" study. J Biopharm Stat. 2019;29(2):378-384. doi: 10.1080/10543406.2018.1535498. Epub 2018 Oct 22. PMID 30346877
- [Background] Dahmane E, Hutson PR, Gobburu JVS. Exposure-Response Analysis to Assess the Concentration-QTc Relationship of Psilocybin/Psilocin. Clin Pharmacol Drug Dev. 2021 Jan;10(1):78-85. doi: 10.1002/cpdd.796. Epub 2020 Apr 6. PMID 32250059
- [Background] Garnett C, Bonate PL, Dang Q, Ferber G, Huang D, Liu J, Mehrotra D, Riley S, Sager P, Tornoe C, Wang Y. Scientific white paper on concentration-QTc modeling. J Pharmacokinet Pharmacodyn. 2018 Jun;45(3):383-397. doi: 10.1007/s10928-017-9558-5. Epub 2017 Dec 5. PMID 29209907
- [Background] Sischka PE, Costa AP, Steffgen G, Schmidt AF. The WHO-5 well-being index - validation based on item response theory and the analysis of measurement invariance across 35 countries. Journal of Affective Disorders Reports. 2020;1(100020).
- See also: ICH Safety Guidelines — https://ich.org/page/safety-guidelines